CLINICAL TRIAL: NCT00996619
Title: Measuring the Spectrum of Tissues During Endoscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: Prof. Arie Orenshtein, Sheba Medical Center
Other Study IDs: SHEBA-7285-09-AO-CTIL
Record Dates: First submitted 2009-09-29; First posted 2009-10-16 (Estimated); Last update posted 2009-10-16 (Estimated); Status verified 2009-10

CONDITIONS: Colon Carcinoma; Colonic Polyps; Intestinal Polyps
MeSH Terms: conditions — Colonic Neoplasms; Colonic Polyps; Intestinal Polyps

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- People undergoing GI tract endoscopy
  Interventions: Procedure: An optical fiber, inside the work channel of an endoscope, is added to the endoscopic examination

INTERVENTIONS:
Procedure: An optical fiber, inside the work channel of an endoscope, is added to the endoscopic examination — An optical fiber, inside the work channel of an endoscope, connected to a spectroscope, enables measuring the spectrum of objects "seen" by the endoscope
  Other Names: The brand of the optical fiber is not relevant

SUMMARY:
Lesions, polyps and other abnormalities in the gastrointestinal (GI) tract have a different composition compared to the normal mucose. The investigators plan to gather spectroscopic information from these features. Characterizing their unique spectrums, may help to enhance the detection and identification of these objects during endoscopy.

ELIGIBILITY:
Inclusion Criteria:

* Adult, independent patients who come to Sheba Hospital's gastro-intestinal clinic for endoscopy and are willing to sign an informed consent

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Independent Adults
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2009-10; Primary Completion 2010-05 (Estimated); Study Completion 2010-05 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Sheba Medical Center, Tel Litwinsky, Israel